CLINICAL TRIAL: NCT05929326
Title: Establishment of Reference Intervals of Complete Blood Count and Coagulation Tests in Pregnant Women at Hung Vuong Hospital
Brief Title: Reference Intervals of Complete Blood Count and Coagulation Tests in Pregnant Women at Hung Vuong Hospital
Status: Completed | Type: Observational
Sponsor: Hung Vuong Hospital (Other)
Collaborators: MITALAB COMPANY LIMITED (Unknown)
Responsible Party: Principal Investigator, Huan Nguyen Pham, Technical supervisor, Hung Vuong Hospital
Other Study IDs: CS/HV/23/13
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related
Keywords: Reference intervals; pregnancy; complete blood count; coagulation tests
MeSH Terms: interventions — Blood Cell Count; Partial Thromboplastin Time

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood samples (2 mL) were collected by plastic whole blood tube with spray-coated K2-EDTA (ethylenediamine tetraacetic acid) Blood samples (2 mL) were collected by plastic whole blood tube with spray-coated Trisodium citrate 3.2%
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First trimester: Pregnant women with gestational age ≤ 13 weeks and 6 days
  Interventions: Diagnostic Test: complete blood count, PT, aPTT, fibrinogen tests
- Second trimester: Pregnant women with gestational age from 14 weeks and 0 days to 27 weeks and 6 days
  Interventions: Diagnostic Test: complete blood count, PT, aPTT, fibrinogen tests
- Third trimester: Pregnant women with gestational age ≥ 28 weeks
  Interventions: Diagnostic Test: complete blood count, PT, aPTT, fibrinogen tests

INTERVENTIONS:
Diagnostic Test: complete blood count, PT, aPTT, fibrinogen tests — Pregnant women who are eligible for the study will have their blood collected to run complete blood count, PT, aPTT, fibrinogen tests

SUMMARY:
Rationale: Pregnancy has major effects on physiology in women. There have been many studies that established reference intervals but none was done in Vietnam. The recommendation by CLSI C28-A3 is that if possible, each laboratory establishes its own reference intervals.

Objective: To establish the reference intervals of complete blood count parameters and Prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen.

Study design: This is a cross-sectional study.

Study population: Pregnant women with no history of disease and normal clinical findings.

DETAILED DESCRIPTION:
Reference intervals (RI) is defined as the central 95% interval of the distribution of values taken from a biological reference population. RI is established for each trimester. The sample needed for each trimester is at least 258 which adds up to 774 when combining three trimesters.

Pregnant women are selected if eligible from obstetrics clinics after history taking and clinical findings. After consent, their blood are then drawn by phlebotomist into an ethylenediamine tetraacetic acid (EDTA) and a trisodium citrate 3.2% blood tube. EDTA samples are run on DxH 900 hematology analyzer, manufactured by Beckman Coulter and citrate samples are run on ACL TOP 550 coagulation analyzer, manufactured by Werfen. The analyzers are verified by laboratory procedure, recommended by Clinical and Laboratory Standards Institute (CLSI) method and quality control is checked before in accordance to the laboratory procedure.

Statistical analysis: Patients were divided into three groups, which are first, second, and third trimester. CLSI EP28-A3c recommended Dixon's D/R ratio outlier test to exclude outliers, where D is the absolute difference between the largest (or smallest) and the second largest (or smallest) observation, and R is the range of all observations. If D is equal to or greater than one-third of R, that observation is considered an outlier and is deleted. After outliers were deleted, the remaining data was tested again for additional outliers until there were no more outliers. A non-parametric method, recommended to establish reference intervals by CLSI EP28-A3c, was used to determine the lower reference limit 2.5th percentile and upper reference limit 97.5th percentile for each group.

Each reference limit was reported along with its 90th confidence interval. Groups were then compared using normal approximation with continuous correction Mann-Whitney U. A two-tailed P-value < 0.05 was considered significant. Statistical analysis was performed using NCSS statistical software (Utah, USA) version 2023

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy

Exclusion Criteria:

* Hypertension, Diabetes, Preeclampsia, Gestational Diabetes, Hemoglobinopathy, Current Infection, Positive Screening for Treponema pallidum, Hepatitis B Virus, HIV, usage of anticoagulant drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women at obstetrics clinics at Hung Vuong Hospital
Sampling Method: Non-Probability Sample
Enrollment: 879 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huan N Pham, Doctor, Principal Investigator — Hung Vuong Hospital
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
data collected will be available when study is completed
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] de Haas S, Ghossein-Doha C, van Kuijk SM, van Drongelen J, Spaanderman ME. Physiological adaptation of maternal plasma volume during pregnancy: a systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2017 Feb;49(2):177-187. doi: 10.1002/uog.17360. PMID 28169502
- [Background] Gong JM, Shen Y, He YX. Reference Intervals of Routine Coagulation Assays During the Pregnancy and Puerperium Period. J Clin Lab Anal. 2016 Nov;30(6):912-917. doi: 10.1002/jcla.21956. Epub 2016 Apr 7. PMID 27061783
- [Background] Jin Y, Lu J, Jin H, Fei C, Xie X, Zhang J. Reference intervals for biochemical, haemostatic and haematological parameters in healthy Chinese women during early and late pregnancy. Clin Chem Lab Med. 2018 May 24;56(6):973-979. doi: 10.1515/cclm-2017-0804. PMID 29303769
- [Background] Cui C, Yang S, Zhang J, Wang G, Huang S, Li A, Zhang Y, Qiao R. Trimester-specific coagulation and anticoagulation reference intervals for healthy pregnancy. Thromb Res. 2017 Aug;156:82-86. doi: 10.1016/j.thromres.2017.05.021. Epub 2017 May 24. PMID 28605659
- [Derived] Pham HN, Huynh NX, Pham PNH, Dang DNY, Cao LT, Huynh DM, Thoi HTT, Le OH, Beaupha SMC. Reference intervals of complete blood count and coagulation tests in Vietnamese pregnant women. BMC Pregnancy Childbirth. 2023 Nov 11;23(1):788. doi: 10.1186/s12884-023-06106-2. PMID 37951881
- See also: Defining, Establishing, and Verifying Reference Intervals in the Clinical Laboratory, 3rd Edition — https://clsi.org/standards/products/method-evaluation/documents/ep28/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Trimester | Second Trimester | Third Trimester
Started | 307 | 279 | 293
Completed | 305 | 276 | 286
Not Completed | 2 | 3 | 7
Not completed — unqualified sample | 2 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- First Trimester: Pregnant women with gestational age ≤ 13 weeks and 6 days
  complete blood count, prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen tests: Pregnant women who are eligible for the study will have their blood collected to run complete blood count, PT, aPTT, fibrinogen tests
- Second Trimester: Pregnant women with gestational age from 14 weeks and 0 days to 27 weeks and 6 days
  complete blood count, prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen tests: Pregnant women who are eligible for the study will have their blood collected to run complete blood count, PT, aPTT, fibrinogen tests
- Third Trimester: Pregnant women with gestational age ≥ 28 weeks
  complete blood count, prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen tests: Pregnant women who are eligible for the study will have their blood collected to run complete blood count, PT, aPTT, fibrinogen tests
- Total: Total of all reporting groups
Arm/Group | First Trimester | Second Trimester | Third Trimester | Total
Number analyzed (Participants) | 305 | 276 | 286 | 867
Age, Customized [Median (Inter-Quartile Range); unit: years] | 28 [25 to 33] | 28 [25 to 32] | 29 [25 to 33] | 29 [25 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 276 | 286 | 867
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Vietnamese | 305 | 276 | 286 | 867
Region of Enrollment [Number; unit: participants]
  Vietnam | 305 | 276 | 286 | 867
Gestational age [Median (Inter-Quartile Range); unit: weeks] | 11 [9 to 12] | 25 [24 to 26] | 37 [36 to 37] | 25 [12 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Trimester Specific Prothrombin Time Reference Interval
Description: Prothrombin time in seconds, measured on ACL TOP 550 coagulation analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: A total of 879 patients were enrolled but 12 patients' samples failed to run, leaving 867 patients. Out of 867 patients, due to unqualified quality, 837 samples were eligible for complete blood count test and 836 samples for coagulation tests
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 288 | 269 | 279
seconds | 11.40 [10.30 to 12.88] | 10.60 [9.80 to 11.60] | 10.40 [9.60 to 11.40]

2. Primary Outcome: Trimester Specific Activated Partial Thromboplastin Time Reference Interval
Description: Activated partial thromboplastin time in seconds, measured on ACL TOP 550 coagulation analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 288 | 269 | 279
seconds | 30.10 [25.40 to 35.50] | 27.90 [24.05 to 33.26] | 27.10 [23.40 to 31.80]

3. Primary Outcome: Trimester Specific Fibrinogen Reference Interval
Description: Fibrinogen in milligram/deciLiter (mg/dL), measured on ACL TOP 550 coagulation analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: mg/dL
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 288 | 269 | 279
mg/dL | 404.56 [280.28 to 559.00] | 450.00 [347.75 to 593.35] | 480.30 [330.28 to 628.56]

4. Primary Outcome: Trimester Specific Hemoglobin Reference Interval
Description: Hemoglobin in gram/deciLiter (g/dL), measured on DxH900 hematology analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: g/dL
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 287 | 273 | 277
g/dL | 12.41 [10.33 to 13.95] | 11.58 [9.71 to 13.17] | 12.11 [9.80 to 13.97]

5. Primary Outcome: Trimester Specific Red Blood Cell Count Reference Interval
Description: Red blood cell count in million cells/μl (M/μl), measured on DxH900 hematology analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: M/μl
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 287 | 273 | 277
M/μl | 4.35 [3.73 to 5.32] | 3.91 [3.33 to 4.98] | 4.18 [3.54 to 4.98]

6. Primary Outcome: Trimester Specific White Blood Cell Count Reference Interval
Description: White blood cell count in thousand cells/μl (K/μl), measured on DxH900 hematology analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: K/μl
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 287 | 273 | 277
K/μl | 9.50 [6.33 to 15.24] | 10.77 [6.99 to 15.55] | 9.48 [6.22 to 14.14]

7. Primary Outcome: Trimester Specific Hematocrit Reference Interval
Description: percentage of hematocrit (%), measured on DxH900 Hematology Analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 287 | 273 | 277
percent | 37.92 [32.22 to 42.23] | 35.13 [30.26 to 40.07] | 37.18 [31.11 to 42.70]

8. Primary Outcome: Trimester Specific Platelet Reference Interval
Description: Platelet in thousand cells/microLiter (K/μl), Measured on DxH900 Hematology Analyzer
Time Frame: Each participant's blood samples are run immediately after phlebotomy within 30 minutes
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: K/μl
Arm/Group | First Trimester | Second Trimester | Third Trimester
Number analyzed (Participants) | 287 | 273 | 277
K/μl | 268.80 [169.66 to 413.88] | 257.70 [172.34 to 372.19] | 249.20 [151.30 to 417.16]

ADVERSE EVENTS:
Time Frame: Adverse events, including all-cause mortality, were not monitored or assessed during the study period. The study was limited to a one-time blood sample collection from each participant between June and August 2023, with no follow-up for adverse events.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored or assessed in this study. The purpose of the study was to evaluate laboratory reference intervals, and no clinical follow-up was performed.
Arm/Group | First Trimester | Second Trimester | Third Trimester
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT05929326/Prot_SAP_000.pdf